CLINICAL TRIAL: NCT04680494
Title: Effect of Acute Physical Exercise on Memory
Acronym: SPEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Igloi Kinga, Senior lecturer, University of Geneva, Switzerland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PB_2017-00360
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Acute Physical Exercise
Keywords: fMRI; BDNF; endocannabinoid; physical exercise
MeSH Terms: conditions — Motor Activity | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: This is a within-subject study, all participants perform all conditions in cross-over randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rest (Experimental): Participants rest quietly for 30 minutes, sitting on a chair. They may read magazines not involving motion-related elements
  Interventions: Other: rest
- Moderate intensity exercise (Experimental): Participants cycle on a cycle ergometer during 30 minutes at 65% of their maximal cardiac frequency
  Interventions: Other: moderate intensity physical exercise
- High intensity exercise (Experimental): Participants cycle on a cycle ergometer during 15 minutes at 75% of their maximal cardiac frequency. This session also includes 3 minutes of warm-up and three minutes of cool down at 50% of their maximal cardiac frequency
  Interventions: Other: high intensity physical exercise

INTERVENTIONS:
Other: moderate intensity physical exercise
  Arms: Moderate intensity exercise
Other: high intensity physical exercise
  Arms: High intensity exercise
Other: rest
  Arms: Rest

SUMMARY:
An increasing amount of studies show the beneficial effect of regular exercise on cognitive and brain functions and especially in the memory domain. Yet little is known of what happens within an acute bout of exercise and whether it would also yield cognitive effects. The literature clearly shows that molecules such as brain derived neurotrophic factor (BDNF) and endocannabinoids (mainly anandamide, AEA) are heavily involved in neural plasticity mechanisms and increase when we exercise hinting at possible mechanisms underlying memory improvement after exercise.

This protocol assesses the effects of acute exercise on associative and motor sequence memory, their underlying neural activations (measured using fMRI) and blood biomarkers (BDNF and AEA). A related aim is to assess the effect of exercise intensity, therefore three exercising conditions (rest, moderate intensity and high intensity) were included. Finally, a 3-month delayed retest visit is also realized to assess effects of acute exercise on long-term memory consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Right-handed,
* Exercising regularly (at least twice per week).
* VO2max comprised between 40ml/kg/min and 65ml/kg/min.

Exclusion Criteria:

- Psychiatric and neurological history

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
cognitive measures - performance | Till the end of the study for each participant, i.e.3 months (long time retest)
  we measure performance during cognitive tasks. Performance is measured as percentage of correct trials, with higher percentages corresponding to better performance - measured in percentages.
cognitive measures - reaction times | Till the end of the study for each participant, i.e.3 months (long time retest)
  we measure reaction times during cognitive tasks. For reaction times, lower measures correspond to faster response times and therefore to better outcome - measured in milliseconds.
BDNF levels | up to 1 hour
  we measure BDNF levels before and after physical exercise and rest, measured in ng/mL of serum.
endocannabinoid levels | up to 1 hour
  we measure endocannabinoid levels before and after physical exercise and rest, measured in ng/mL of plasma.
brain activations | up to 1 hour
  we measure brain activations using fMRI during cognitive tasks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marin Bosch B, Bringard A, Logrieco MG, Lauer E, Imobersteg N, Thomas A, Ferretti G, Schwartz S, Igloi K. Effect of acute physical exercise on motor sequence memory. Sci Rep. 2020 Sep 18;10(1):15322. doi: 10.1038/s41598-020-72108-1. PMID 32948800